CLINICAL TRIAL: NCT04621929
Title: Phentermine/tOpiramate to eND Obesity and Uric Acid Stones Trial (POuND OUT)
Brief Title: Phentermine/Topiramate for Uric Acid Stones
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202001895-A-N; 1R21DK122317-01A1 (NIH)
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Uric Acid Stones; Type 2 Diabetes Mellitus in Obese; Pre-Diabetes
MeSH Terms: conditions — Obesity; Glucose Intolerance | interventions — Phentermine; Topiramate; Qsymia; Allopurinol; Diet

STUDY DESIGN:
Intervention Model Description: 2:1 ratio block site of 6
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Allocated to intervention/treatment (Experimental): Daily phentermine/topiramate x 18 months
  Interventions: Drug: Phentermine / Topiramate Oral Product
- Allocated to pragmatic control (Active Comparator): Remain on their current regimen
  Interventions: Combination Product: Citrate Salts, Allopurinol, Diet

INTERVENTIONS:
Drug: Phentermine / Topiramate Oral Product — All participants in the experimental group will receive oral generic tablet phentermine (18.75 or 37.5 mg dose) and topiramate (daily 100 mg or 150 mg dose)
  Other Names: Duromine; Adipex-P; Lomaira; Suprenza; Trokendi XR; Topamax; Qudexy XR; Eprontia; Qsymia
  Arms: Allocated to intervention/treatment
Combination Product: Citrate Salts, Allopurinol, Diet — Control participants will complete initial visit requirements and study enrollment and will be maintained on their current therapy.
  Arms: Allocated to pragmatic control

SUMMARY:
The investigator proposes an 18 month, feasibility pilot study, randomizing obese and diabetic individuals with pure uric acid nephrolithiasis (UAN) or mixed calcium oxalate (CO) UAN to either phentermine/topiramate or a pragmatic control group who will remain on their standard medication regimen (citrate salts, allopurinol, diet, etc.).

DETAILED DESCRIPTION:
Mounting evidence indicates that obesity, diabetes mellitus, and kidney stones are inter-connected diseases, particularly uric acid nephrolithiasis (UAN) with or without components of calcium oxalate (CO). Obese or overweight diabetics have a six-fold increased risk to develop UAN/COUAN due to the inability to properly add buffer (ammonium) to urine. Of the FDA approved drugs in the weight loss market, the combination medication phentermine/ topiramate is the most effective and has a unique side effect of alkalinizing the urine (making it less acidic). The hypothesize of this project is that treatment of obese, diabetic patients with phentermine/topiramate will reduce the incidence of UAN/COUAN by 1) direct urinary alkalinization and 2) weight loss. Weight loss will indirectly improve urinary buffering ability through improvement in insulin sensitivity and will decrease renal oxidative stress. The investigative team proposes an 18 month, feasibility pilot study, randomizing 30 obese and diabetic individuals with UAN/COUAN to either phentermine/topiramate (n=20) or a pragmatic control group (n=10) who would remain on standard medication regimen (citrate salts, allopurinol, diet, etc).

ELIGIBILITY:
Inclusion Criteria:

* have recurrent pure uric acid nephrolithiasis (UAN) or mixed calcium oxalate (CO)/UAN. Recurrent stone disease is defined as at least two spontaneous kidney stone passages, two previous kidney stone procedures, or one previous stone passage and one previous procedure. Pure UAN is defined as at least one previous stone analysis demonstrating 100% uric acid mineral content. Mixed COUAN will be defined as at least one previous stone analysis with any mix of uric acid ≥80% and ≤20% calcium oxalate. If participant has more than one stone analysis, the most recent will be considered the current stone type.
* have obesity, defined as BMI > 30 kg/m2.
* have type 2 diabetes mellitus or pre-diabetes, defined as previously diagnosed by laboratory testing (hemoglobin A1c, fasting plasma glucose, or oral glucose tolerance test) or as demonstrated by use of anti-hyperglycemic medications or insulin.
* have at least one 24-hour urine study off medications demonstrating urine pH < 5.8 or a study 24-hr urine demonstrating urine pH < 5.8

Exclusion Criteria:

* contraindications to topiramate, including: recurrent major depression, current substantial depressive symptoms, uncontrolled depression by PHQ 9 score >= 10, history of suicidal ideation or behavior with intent to act (versus exclude those with depression); current pregnancy or attempting to conceive; pre-existing chronic kidney disease with eGFR < 60 at time of enrollment; active cancer or active treatment for cancer (chemotherapy, radiation); and non-ambulatory.
* contraindications to phentermine, including: unstable cardiovascular disease defined as decompensated heart failure, unstable angina, atrial fibrillation, uncontrolled blood pressure (>160 systolic), hyperthyroidism; monoamine oxidase inhibitor use; current history of drug or alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Canales, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allocated to Intervention/Treatment | Allocated to Pragmatic Control
Started | 13 | 6
Completed | 10 | 5
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allocated to Intervention/Treatment | Allocated to Pragmatic Control | Total
Number analyzed (Participants) | 13 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.80 (9.5) | 69.20 (6.4) | 64 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 6 | 17
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Kidney Stone Size (mm^3) Determined by Non-contrast CAT Scan
Description: Stone perimeter within each cut of CT image was outlined using semiautomated volume tool (region of interest pen tool, CT software "Visage Imaging") and tallied to calculate stone volume (mm^3) for each individual stone and recorded from right and left kidney from all study participants at baseline CT and at end of study CT (18 months)
Time Frame: Baseline, 18 months
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Allocated to Intervention/Treatment | Allocated to Pragmatic Control
Number analyzed (Participants) | 13 | 6
mm^3
  Baseline | 6540 (10430) | 4650 (6064)
  End of Study (18 months) | 3120 (5158) | 5041 (7043)

2. Secondary Outcome: Weight (kg)
Description: total weight (baseline and end of study)
Time Frame: Baseline, 18 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Allocated to Intervention/Treatment | Allocated to Pragmatic Control
Number analyzed (Participants) | 13 | 6
kg
  Baseline | 121.4 (24) | 101.2 (23)
  End of Study (18 months) | 111.2 (24) | 104.1 (26)

3. Secondary Outcome: Urinary pH Parameters
Description: urine pH (baseline and end of study). The pH scale ranges from 0 to 14. A pH of 7 is neutral. A pH less than 7 is acidic. A pH greater than 7 is basic.
Time Frame: Baseline, 18 months
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Allocated to Intervention/Treatment | Allocated to Pragmatic Control
Number analyzed (Participants) | 13 | 6
unitless
  Baseline | 5.3 (0.2) | 5.3 (0.2)
  End of Study (18 months) | 6.2 (0.5) | 5.5 (0.5)

4. Secondary Outcome: %Hemoglobin A1c
Description: %A1c (baseline and end of study)
Time Frame: Baseline, 18 months
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Allocated to Intervention/Treatment | Allocated to Pragmatic Control
Number analyzed (Participants) | 13 | 6
percentage of glycated hemoglobin
  Baseline | 6.6 (1.4) | 6.2 (0.9)
  End of Study (18 months) | 6.4 (1.5) | 6.7 (1.5)

5. Secondary Outcome: Urinary Citrate Parameters
Description: urinary citrate (baseline and end of study)
Time Frame: Baseline, 18 months
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Allocated to Intervention/Treatment | Allocated to Pragmatic Control
Number analyzed (Participants) | 13 | 6
mg/day
  Baseline | 634 (289) | 673 (526)
  End of Study | 309 (81) | 951 (782)

6. Secondary Outcome: Urinary Calcium Parameters
Description: urinary calcium (baseline and end of study)
Time Frame: Baseline, 18 months
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Allocated to Intervention/Treatment | Allocated to Pragmatic Control
Number analyzed (Participants) | 13 | 6
mg/day
  Baseline | 172 (58) | 154 (95)
  End of Study (18 months) | 224 (45) | 167 (122)

7. Secondary Outcome: Urinary Uric Acid Supersaturation (SS)
Description: Urinary uric acid SS (before and end of study). Urinary Uric Acid Supersaturation (SS) is not measured in a specific unit, as it is a ratio. Result below 1: The urine is undersaturated, meaning that crystals are more likely to dissolve than form. Result equal to 1: The urine is in equilibrium with uric acid, so crystals will not grow or shrink. Result above 1: The urine is supersaturated, and the risk for crystals to form and grow is increased. A higher value indicates a greater risk.
Time Frame: Baseline, 18 months
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Allocated to Intervention/Treatment | Allocated to Pragmatic Control
Number analyzed (Participants) | 13 | 6
unitless
  Baseline | 2.2 (1.1) | 2.4 (1.0)
  End of Study (18 months) | 0.7 (1.1) | 1.8 (1.1)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Allocated to Intervention/Treatment | Allocated to Pragmatic Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6
Other Adverse Events (participants affected / at risk) | 12/13 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allocated to Intervention/Treatment (N=13) | Allocated to Pragmatic Control (N=6)
Kidney Stone Passage (Renal and urinary disorders) | 3 (3) | 3 (3)
Kidney Stone Procedure (Renal and urinary disorders) | 0 (0) | 2 (2)
Dizziness (General disorders) | 1 (1) | 0 (0)
Dysgeusia (General disorders) | 1 (1) | 0 (0)
Erectile Dysfunction (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Menstrual Cycle Irregularity (Reproductive system and breast disorders) | 1 (1) | 0 (0)
New Onset Artrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bladder Stone Surgery (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT04621929/Prot_001.pdf
  • Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT04621929/SAP_002.pdf
  • Informed Consent Form (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT04621929/ICF_000.pdf